CLINICAL TRIAL: NCT06526455
Title: Efficacy and Safety of Vonorasan Versus Esomeprazole in the Treatment of Ulcers After Endoscopic Submucosal Dissection (ESD): a Multicentre, Parallel-design, Double-blind, Randomised Controlled Study
Brief Title: Efficacy and Safety of Vonorasan Versus Esomeprazole in the Treatment of Ulcers After Endoscopic Submucosal Dissection
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shicai Ye (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Maoming People's Hospital (Other); Yellow River Sanmenxia hospital (Unknown)
Responsible Party: Sponsor-Investigator, Shicai Ye, chief physician, Affiliated Hospital of Guangdong Medical University
Organization: Affiliated Hospital of Guangdong Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PJKT2024-109
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Ulcers, Gastric
MeSH Terms: conditions — Stomach Ulcer | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Vonorasan、tablet、20mg、qd、Days 3 to 56
  Interventions: Drug: Vonoprazan
- Control group (Active Comparator): Esomeprazole 、tablet、20mg、Days 3 to 56
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan — oral drug 3-56 days after ESD.
  Arms: Treatment group
Drug: Esomeprazole — oral drug 3-56 days after ESD.
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to find out the effectiveness of voronasan in combination with aluminum phosphate gel in the treatment of post-operative ESD ulcers. It will also find out about the safety of vunorasan in combination with aluminum phosphate gel. The main questions it aims to answer are:

1. Do vonorasan in combination with aluminum phosphate gel clinically effective in the treatment of post-operative ESD ulcers?
2. What medical problems do participants have when taking drug vonorasan in combination with aluminum phosphate gel? Researchers compared the drug voransen in combination with aluminum phosphate gel to esomeprazole in combination with aluminum phosphate gel to see if voransen in combination with aluminum phosphate gel worked better for post-operative ESD ulcers.

Participants will:

Intravenous lansoprazole 1-3 days after ESD and oral voronasan combined with aluminum phosphate gel or esomeprazole combined with aluminum phosphate gel 3-56 days after ESD.

Record their symptoms, endoscopic ulcer grading, ulcer size and Calculate ulcer healing rate at weeks 2 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Meets surgical indications for ESD
* Age 18-70 years, regardless of gender
* Normal coagulation
* ESD Postoperative ulcers ≤3cm
* Voluntary participation in the study

Exclusion Criteria:

* Patients with severe complications or failure to achieve curative resection after gastric ESD surgery need supplementary surgery
* Women who are pregnant or breastfeeding, or who may conceive during clinical trials
* The patient has other serious organic diseases that affect the evaluation of the study, such as severe liver disease, heart disease, renal disease, malignant neoplasm and alcoholism
* Patients who need to take antiplatelet and NSAIDS drugs for a long period of time
* Co-administration of unspecified anti-ulcer drugs during the trial period;Allergic reactions to vornoxan, aluminium phosphate gel or esomeprazole
* Patients with no capacity for autonomous behaviors, unable to correctly express their main complaint, such as those with mental illness, severe neurosis, and unable to cooperate with this experiment
* ESD Postoperative ulcers >3cm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of ulcer reduction | 2nd and 8th week post-dose
  Ulcer area = maximum diameter of the ulcer * perpendicular line of the maximum diameter (mm2) The rate of ulcer reduction at 2 weeks = [(area of the initial ulcer - area of the ulcer at 2 weeks)/area of the initial ulcer]*100% The rate of ulcer reduction at 8 weeks = [ (area of the initial ulcer - area of the ulcer at 8 weeks)/area of the initial ulcer]*100% Ulcer area = maximum diameter of the ulcer * perpendicular line of the maximum diameter (mm2) The rate of ulcer reduction at 2 weeks = [(area of the initial ulcer - area of the ulcer at 2 weeks)/area of the initial ulcer]*100% The rate of ulcer reduction at 8 weeks = [ (area of the initial ulcer - area of the ulcer at 8 weeks)/area of the initial ulcer]*100%

SECONDARY OUTCOMES:
Size of ulcer | 2nd and 8th week post-dose
  Ulcer area = maximum diameter of the ulcer * perpendicular line of the maximum diameter (mm2)
Rate of ulcer healing | 2nd and 8th week post-dose
  Healing rate = number of cases with scarring/total number of cases × 100 per cent
Rate of bumpy | 2nd and 8th week post-dose
  Rate of bumpy= number of cases that have occurred/total number of cases × 100 per cent
Quality of ulcer healing | 2nd and 8th week post-dose
  Scoring using the Ulcer Healing Scoring Scale，the highest score is 3 and the lowest is 1, with higher scores indicating better ulcer healing
Rate of delayed hemorrhage | 2th week post-dose
  Rate of delayed hemorrhage=Number of haemorrhages/total
Postoperative symptom relief rate | 2th week post-dose
  Number of persons in remission/total

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Yellow River Sanmenxia Hospital, Sanmenxia, Henan